CLINICAL TRIAL: NCT06019520
Title: Role of N-Acetylcysteine for Prevention of Cisplatin-induced Nephrotoxicity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FUI/CTR/2023/14
Record Dates: First submitted 2023-08-18; First posted 2023-08-31 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Drug Toxicity
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions | interventions — Acetylcysteine; Drug Therapy

STUDY DESIGN:
Intervention Model Description: It will be a two-arm study with 35 patients in each arm. After taking informed consent, a total of 70 patients will be enrolled. The patients will be enrolled by convenience nonprobability sampling technique. Then they will be randomized to the N-Acetylcysteine plus chemotherapy and chemotherapy-alone arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cisplatin group (Active Comparator): This group of Patients will receive Cisplatin-base chemotherapy as per the designated schedule, alongside standard hydration protocol
  Interventions: Drug: Chemotherapy
- N-acetylcysteine group (Experimental): Patients in the NAC arm to be given N-acetylcysteine 1200 mg/day starting 12 hrs before till 6 days after Cisplatin-based chemotherapy administration. Hydration according to standard hydration protocol will be given.
  Interventions: Drug: N-Acetylcysteine; Drug: Chemotherapy

INTERVENTIONS:
Drug: N-Acetylcysteine — Patients in the NAC arm will receive1200 mg of NAC (water-soluble granule Preparation) administered orally once daily at night for 7 consecutive days (1 days before chemotherapy, on the day of chemotherapy, and 5 days after chemotherapy) in each cycle of chemotherapy.
  Arms: N-acetylcysteine group
Drug: Chemotherapy — Cisplatin-base chemotherapy as per the designated schedule, alongside standard hydration protocol.

SUMMARY:
Cisplatin is one of the first-line drugs used against many malignancies, such as lung cancer, head and neck cancer, esophageal cancer, gastric cancer, colorectal cancer, urothelial cancer, bladder cancer and testicular cancer. The usage of Cisplatin is limited by its severe nephrotoxicity, which particularly affects the proximal tubule epithelial cells (PTEC).Several studies suggest role of NAC in ameliorating Cisplatin induced nephrotoxicity, although definitive data is lacking. N-Acetylcysteine (NAC) is a thiol-containing antioxidant, which not only acts as a precursor of glutathione but also as a direct antioxidant .There are multiple postulated mechanisms for NAC's nephroprotection. NAC is a low-cost, easily available drug with a very good safety profile and therefore can be added as a support medication during treatment with cisplatin. The investigators plan to administer 1200 mg oral NAC 12 hours before chemotherapy and then daily at night for the subsequent 6 days, with an objective to ascertain its nephroprotective role in population receiving Cisplatin/-based chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult female outpatients with non-hematological malignancies (Breast, ovary and head and neck squamous cell carcinomas)
* Having Eastern Cooperative Oncology Group(ECOG) Performance Status ≤2 who had never received platinum based Chemotherapy in past and were now scheduled to receive high-dose cisplatin chemotherapy.
* Patients were required to have estimated glomerular filtration rate (GFR)(according to Cockcroft-Gault formula) ≥ 60 ml/min at start of chemotherapy regimen with normal Blood Counts, Liver, and kidney function tests

Exclusion Criteria:

* Patients who had poor performance status i.e., ECOG Performance Status 3 or 4
* Who declined to participate at any time during the course of the study
* Patients having hepatic failure (Liver Function tests >3 times of upper limit normal)
* Patients who did not tolerate the use of NAC or were administered the drug <70% of the time
* Patient who were receiving concurrent nephrotoxic drugs, or having history of Hypersensitivity to N-Acetyl cysteine.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The study includes adult female outpatients with non-hematological malignancies
Enrollment: 70 (Estimated)
Dates: Start 2023-08-09 (Actual); Primary Completion 2024-02-09 (Estimated); Study Completion 2024-03-09 (Estimated)

PRIMARY OUTCOMES:
Serum creatinine of participant | 18 weeks
  Blood samples collected and measured in laboratory with the unit mg/dL
Creatinine clearance of participant | 18 weeks
  It will be calculated using Cockroft-Gault formula , unit ml/min
Estimation of Acute kidney injury to participant | 18 weeks
  Acute kidney injury will be assessed by RIFLE criteria that will be calculated for patients
Blood urea nitrogen of participant | 18 weeks
  Blood samples collected and measured in laboratory with the unit mg/dl

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Oncology department, Fauji Foundation Hospital, Rawalpindi, Punjab Province, Pakistan